CLINICAL TRIAL: NCT05527444
Title: The Clinical Efficacy and the Changes of Immune Cells Subsets With Bioagents in Ankylosing Spondylitis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: effecacy of bioagents-AS QiluH
Record Dates: First submitted 2022-05-06; First posted 2022-09-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Ankylosing Spondylitis
Keywords: secukinumab; adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab; Adalimumab; Anti-Inflammatory Agents, Non-Steroidal; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized-SEC group (Experimental): actived AS patients naïve to ADA and SEC
  Interventions: Drug: Secukinumab 150 mg/ml; Drug: NSAID; Drug: Thalidomide Pill
- Randomized-ADA group (Experimental): actived AS patients naïve to ADA and SEC
  Interventions: Drug: Adalimumab Ab; Drug: NSAID; Drug: Thalidomide Pill
- Non-Randomized-SEC group (Experimental): AS patients who previously had inadequate response to ADA
  Interventions: Drug: Secukinumab 150 mg/ml; Drug: NSAID; Drug: Thalidomide Pill
- Non-Randomized-ADA group (Experimental): AS patients who previously had inadequate response to SEC
  Interventions: Drug: Adalimumab Ab; Drug: NSAID; Drug: Thalidomide Pill

INTERVENTIONS:
Drug: Secukinumab 150 mg/ml — Secukinumab 150 mg will be administered at Baseline, Week 1, 2, 3, 4, 6, 8 followed by dosing every 4 weeks until Week 24
  Other Names: Secukinumab
  Arms: Non-Randomized-SEC group; Randomized-SEC group
Drug: Adalimumab Ab — adalimumab biosimilar 40 mg will be administered at Baseline followed by dosing every 2 weeks until Week 24
  Other Names: Adalimumab
  Arms: Non-Randomized-ADA group; Randomized-ADA group
Drug: NSAID — stable dose
Drug: Thalidomide Pill — If patients have inadequate response to bioagents, thalidomide 50 mg will be administered at 12 week followed by dosing everyday until Week 24.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy, safety and immunological changes of secukinumab(sec) compared to adalimumab(ada) in patients with active ankylosing spondylitis(AS), who previously have an inadequate response to non-steroidal anti-inflammatory drugs (NSAIDs) or bioagents.

DETAILED DESCRIPTION:
Biologic naïve participants will be randomly assigned in a 2:1 ratio to receive secukinumab or adalimumab for 24 weeks. Participants with a history of an inadequate response to secukinumab or adalimumab, will be treated with the alternative drug (adalimumab or secukinumab) for 24 weeks. The disease activity and index of inmunology will be evaluated at weeks 0, 12, 24 up to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet modified New York 1984 criteria for ankylosing spondylitis；
2. Age ≥18 years and ≤ 65 years；
3. ASDAS ≥ 1.3；
4. Concomitant drugs: use stable doses of NSAIDs alone for at least 4 weeks before the baseline period, stop other oral drugs such as methotrexate (MTX), sulfasalazine (SASP), glucocorticoids. Glucocorticoids can be injected locally after 12 weeks, NSAIDs keep stable for 12 weeks；
5. Willing to participate in this study, willing to medication and follow-up according to the treatment plan, and sign the informed consent.

Exclusion Criteria:

1. Patients with severe infections, tumors and damage to vital organs:

   * Platelet counts(PLT) <80 x 10^9 / L, or white blood cell (WBC) <3 x10^9 / L;
   * Propionate acid aminotransferase (ALT) or aspartate aminotransferase(AST) is two times higher than the upper limit of normal;
   * Renal insufficiency: serum Cr ≥ 176 umol / L;
   * Pregnant or nursing women (breastfeeding) ;
   * Patients has a history of malignancy (cure time in less than 5 years);
   * Patients with severe or poorly controlled hypertension, diabetes or cardiac dysfunction;
2. Patients with current or previous Crohn's disease;
3. Patients with current ulcerative colitis requiring immunosuppressive therapy;
4. Any active infection Active viral hepatitis includes hepatitis B virus (HBV), hepatitis C virus (HCV), human papillomavirus (HPV). Active infections include small intestine herpes zoster virus (VZV), human immunodeficiency virus (HIV), syphilis or tuberculosis;
5. Patients who have received live vaccines within 4 weeks before randomization or plan to receive live vaccines during the trial;
6. Patients who had inadequate response, intolerance or contraindication for both adalimumab and secukinumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline and Week 12
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe]) Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity]) Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe]) Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours]) High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.

SECONDARY OUTCOMES:
Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 20 Response | Baseline and Week 12, 24, 96
  ASAS 20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline and Week 24, 96
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe]) Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity]) Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe]) Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours]) High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 40 Response | Baseline and Week 12, 24, 96
  ASAS 40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response | Baseline and Week 12, 24, 96
  The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from Baseline in BASDAI score.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline and Week 12, 24, 96
  The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMI[Lin]) | Baseline and Week 12, 24, 96
  The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  cervical rotation (measured in degrees), tragus to wall distance (in centimeters [cm]) lumbar side flexion (in cm), lumbar flexion (modified Schober's) (in cm) and intermalleolar distance (in cm). Each measurement is converted to a linear score between 0 and 10. The total BASMI score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Change From Baseline in ASAS Health Index (HI) | Baseline and Week 12, 24, 96
  The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. Each of the 17 questions is answered by the participant as "I agree" (score = 1) or "I disagree" (score = 0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, where a higher score indicates a worse health status. A negative change from Baseline indicates improvement.
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) | Baseline and Week 12, 24, 96
  Change from Baseline in ESR, ESR will be measured with blood samples.
Change From Baseline in C-reactive Protein (CRP) | Baseline and Week 12, 24, 96
  Change from Baseline in C-reactive Protein (CRP), a component index of ASDAS will be measured with blood samples.
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | Baseline and Week 12, 24, 96
  The MASES evaluation was conducted to assess the presence or absence of enthesitis (inflammation of the entheses, or sites where tendons or ligaments insert into the bone) at 13 different sites (first costochondral joint left/right, seventh costochondral joint left/right, posterior superior iliac spine left/right, anterior superior iliac spine left/right, iliac crest left/right, fifth lumbar spinous process, and proximal insertion of Achilles tendon left/right. Each site was scored for presence (1) or absence (0) of enthesitis. The MASES is the sum of the 13 site scores, and ranges from 0 to 13, with higher scores indicating more inflammation of the entheses.
modiifed stoke ankylosing spondylitis spine score (mSASSS) | Baseline and Week 96
  modiifed stoke ankylosing spondylitis spine score ( range 0-72), a system for grading and evaluating cervical spine, lumbar spine, sacroiliac joint and hip joint by X-ray.
Dynamics of T Cell subset | Baseline and Baseline and Week 12, 24
  T cell subsets, including cytotoxic T (Tc) cells, helper T (Th) cells

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiaoyun, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No